CLINICAL TRIAL: NCT03722212
Title: Evaluation of METAglut1 Diagnostic Test Performances in Patients With a Clinical Suspicion of GLUT1 Deficiency Syndrome
Brief Title: Early Diagnosis of the GLUT1 Deficiency Syndrome With a Blood Based Test
Acronym: METAglut1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: METAFORA biosystems (Industry)
Collaborators: European Commission (Other); Assistance Publique - Hôpitaux de Paris (Other); Cemka-Eval (Other); Ministry for Health and Solidarity, France (Other Government); French National Authority for Health (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A01473-50
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-08

CONDITIONS: Glut1 Deficiency Syndrome; De Vivo Disease; Seizures; Movement Disorders; Intellectual Disability; Ataxia
Keywords: Glut1 Deficiency Syndrome; Glut1DS
MeSH Terms: conditions — Glut1 Deficiency Syndrome; Seizures; Movement Disorders; Intellectual Disability; Ataxia

STUDY DESIGN:
Intervention Model Description: The METAglut1 test is performed on each patient, in parallel and blindly of the reference diagnostic strategy which is performed through the current practice (lumbar puncture (LP) performed in the fasting state with glycemia measured right before LP, followed by genetic analyses (targeted slc2a1 analysis or gene panels or whole exome sequencing).
Masking Description: The METAglut1 test is performed blindly of the reference strategy. METAglut1's result masking is maintained for the investigator on the one hand, and the glycorrhachia value masking is maintained for the centralized testing laboratory in charge of METAglut1 on the other hand.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective patients (Other): The METAglut1 test is performed on all patients included in the study. In parallel, patients included prospectively (based on a clinical suspicion) benefit from the reference diagnostic strategy through the current practice, starting with a lumbar puncture for glycorrhachia dosage.
  Interventions: Diagnostic Test: METAglut1
- Retrospective patients (Other): Patients with confirmed Glut1DS diagnosis Already diagnosed patients are included retrospectively as well as patients with pending diagnosis at inclusion (inconsistent biological or genetic data).
  Interventions: Diagnostic Test: METAglut1

INTERVENTIONS:
Diagnostic Test: METAglut1 — A blood draw is performed on each patient for the METAglut1 test, and sent to Laboratoire CERBA, Saint-Ouen l'Aumône, France, for sample analysis.

SUMMARY:
The study aims at validating the diagnostic performances of the METAglut1, a blood in vitro diagnostic test, for the simple and early diagnosis of the Glut1 deficiency syndrome (Glut1DS, or De Vivo disease).

The blood test will be carried out prospectively on patients presenting with a clinical suspicion of Glut1DS, blindly from the reference strategy, which consists in a lumbar puncture for glycorrhachia measurement, completed by a molecular analysis.

The study will be conducted in more than 40 centers in France on up to 3,000 patients for 2 years.

DETAILED DESCRIPTION:
The Glut1 Deficiency Syndrome (Glut1DS) is a debilitating, proteiform neurometabolic disorder caused by an impairment in the glucose transporter Glut1 at the cell surface. Patients suffer from seizures, movement disorders and intellectual disabilities. A timely diagnosis is of prime importance as this haploinsufficiency can be improved by the so-called ketogenic diet.

By diagnosing Glut1DS early, based on symptoms associated with Glut1DS, healthcare providers can prescribe the Keto diet therapy early in the disease progression, which could prevent impairment of central nervous system function caused by the disease. Therefore, an early diagnosis of Glut1DS for its treatment is crucial.

Currently, the disease is very difficult to diagnose correctly and in a timely manner. The current diagnosis practice requires a lumbar puncture in order to determine if hypoglycorrhachia occurs. The diagnosis result is then supported by the detection of a heterozygous pathogenic variant in slc2a1 gene. This diagnosis procedure is time consuming, expensive, and requires a geneticist's data interpretation. Currently, ketogenic diet therapy is the most efficient therapy for Glut1DS.

METAglut1 is a first-in-kind IVD device used to aid in the diagnosis of the Glut1 Deficiency Syndrome (Glut1DS) by quantifying the cell surface expression level of the glucose transporter 1 (Glut1) on circulating human red blood cells. The METAglut1 IVD is primarily intended for use in pediatric patients older than 3 months, of both sexes, of any ethnic origin. The METAglut1 IVD may also be used to aid in the diagnosis of Glut1DS in adults with late onset symptoms.

The METAglut1 IVD is authorized for marketing in the European Union pursuant to the CE mark and is currently being distributed in France.

The study aims to validate the diagnostic performances of METAglut1. It will last for 2 years, more than 40 centers will participate in the study across France. Up to 3,000 patients with symptoms compatible with Glut1DS will be included prospectively; each of them will be tested for METAglut1, in parallel and blindly of the reference strategy. The METAglut1 test is performed by Laboratoire CERBA (Saint-Ouen l'Aumône, France). A retrospective cohort of already diagnosed patients will also be analyzed to add more data. Concordance analysis with the glycorrhachia, the first biochemical dosage involved in the reference strategy, will be performed, and overall diagnostic performances of METAglut1 calculated.

Before to start analysis, a thorough data management plan was implemented with on-site monitoring, automated controls of eCRF and recoding after queries and data reviewing.

ELIGIBILITY:
Prospective patients - Inclusion Criteria:

* Clinical suspicion of the GLUT1 Deficiency Syndrome

Retrospective patients - Inclusion Criteria:

* Patients with confirmed Glut1DS diagnosis
* Patients with pending diagnosis at inclusion (inconsistent biological or genetic data)

Exclusion Criteria (for both cohorts):

* Patients under 3 months of age
* Sickle cell disease S/S
* Abnormal imaging

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Concordance analysis between METAglut1 and glycorrhachia | Up to 6 months
  This analysis will be performed on patients with a diagnosis of certainty, either positive or negative, in the prospective cohort. For this analysis two subgroups are distinguished:
  * Patients with lumbar puncture, molecular analysis of the slc2a1 gene and METAglut1 testing.
  * Patients with at least lumbar puncture and METAglut1 testing.

SECONDARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive values of METAglut1 | Up to 6 months
  These analysis will be performed on patients with a diagnosis of certainty in the prospective cohort. For this analysis two subgroups are distinguished:.
  * Patients with at least lumbar puncture and METAglut1 testing.
  * Patients with at least molecular analysis of the slc2a1 gene and METAglut1 testing.

OTHER OUTCOMES:
Sensitivity, specificity of METAglut1 | Up to 6 moths
  These analysis will be performed on patients with a diagnosis of certainty in the retrospective cohort and cumulated cohort (prospective and retrospective). For this analysis two subgroups are distinguished:.
  * Patients with at least lumbar puncture and METAglut1 testing.
  * Patients with at least molecular analysis of the slc2a1 gene and METAglut1 testing.
Concordance analysis between METAglut1 and glycorrhachia | Up to 6 months
  This analysis will be performed on patients with at least lumbar puncture and METAglut1 testing and with a diagnosis of certainty, either positive or negative, in the cumulative cohort (prospective and retrospective).
Sensitivity analysis with optimized threshold of positivity of the METAglut1™ assay | Up to 6 months
  In a sensitivity analysis, the threshold of positivity of the METAglut1™ assay will vary between 75% and 80% and performances calculations will be reported for this variation.
Time to diagnosis | Up to 6 months
  The time between clinical suspicion of Glut1DS and diagnosis will be calculated and compared between different diagnostic strategies
Health technology assessment | Up to 2 years
  Health technology assessment will be performed on patients included in the study

CONTACTS AND LOCATIONS:
Overall Officials: Fanny Mochel, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (28):
- France (28):
  - Hôpital Larrey- CHU Angers, Angers
  - Hôpital Saint Léon, Bayonne
  - Hôpital Jean Verdier- APHP, Bondy
  - Centre hospitalier Pellegrin_ CHU Bordeaux, Bordeaux
  - Hôpital Femme Mere enfant- CHU de Lyon, Bron
  - Hospices Civils de Lyon_CHU Lyon, Bron
  - Hôpital d'Estaing- CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon Bourgogne, Dijon
  - Hôpital Raymond Poincaré- APHP, Garches
  - Hôpital Nord_CHU Grenoble, La Tronche
  - Hôpital Jeanne de Flandre _CHRU Lille, Lille
  - Hôpital de la mère et de l'enfant- CHU Limoges, Limoges
  - Hôpital La Timone Enfant- APHM, Marseille
  - CHR Metz-Thionville, Metz
  - Hôpital Gui de Chauliac- CHU Montpellier, Montpellier
  - Hôpital Mère-Enfant_ CHU de Nantes, Nantes
  - Hôpital la Pitié-Salpêtrière-APHP, Paris
  - Hôpital Necker- APHP, Paris
  - Hôpital Robert Debré- APHP, Paris
  - Hôpital Trousseau- APHP, Paris
  - Hôpital Bicêtre- APHP, Paris
  - Hôpital Sud de Rennes- CHU Rennes, Rennes
  - Hôpital de Saint-Nazaire, Saint-Nazaire
  - Hôpital Nord, CHU Saint-Etienne, Saint-Priest-en-Jarez
  - Hôpital de Hautepierre- CHU Strasbourg, Strasbourg
  - Hôpital de Tarbes - CH Bigorre, Tarbes
  - Hôpital des Enfants- CHU Toulouse, Toulouse
  - Hôpital de Clocheville_ CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding authors on reasonable request. Permissions are required to gain access to the data resources, subject to successful registration and application process.

REFERENCES:
- [Background] Gras D, Cousin C, Kappeler C, Fung CW, Auvin S, Essid N, Chung BH, Da Costa L, Hainque E, Luton MP, Petit V, Vuillaumier-Barrot S, Boespflug-Tanguy O, Roze E, Mochel F. A simple blood test expedites the diagnosis of glucose transporter type 1 deficiency syndrome. Ann Neurol. 2017 Jul;82(1):133-138. doi: 10.1002/ana.24970. PMID 28556183
- See also: METAglut1's project website — http://www.metafora-biosystems.com